CLINICAL TRIAL: NCT07390734
Title: Patient Specific 3d Titanium Plate Versus Standard Two Mini Plates in the Fixation of Mandibular Angle Fractures (a Randomized Controlled Clinical Trial)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1023-01/2025
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Mandibular Angle Fracture
Keywords: three dimensional plates; mandibular angle fracture; patient specific plate

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Masking Description: Participants complying with the inclusion criteria will be randomly assigned using a computer-generated list of random numbers to one of the two arms. Allocation will be performed by a trial independent individual and the allocation ratio is intended to be equal. Allocation will be in equal blocks to ensure that the study groups have equal number of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with recent mandibular angle fractures managed with custom-made 3D titanium plates (Experimental): patients that will undergo internal fixation with custom-made 3D titanium plates through intaoral and transbuccal approach .
  Interventions: Device: custom-made 3D titanium plates
- patients with recent mandibular angle fractures managed with standared two mini plates (Experimental): patient that will undergo internal fixation with standared two mini plates through intaoral and transbuccal approach.
  Interventions: Device: standared two mini plates

INTERVENTIONS:
Device: custom-made 3D titanium plates — custom-made 3D titanium plates through intaoral and transbuccal approach .
  Arms: patients with recent mandibular angle fractures managed with custom-made 3D titanium plates
Device: standared two mini plates — internal fixation with standared two mini plates through intaoral and transbuccal approach.
  Arms: patients with recent mandibular angle fractures managed with standared two mini plates

SUMMARY:
To compare the effectiveness of custom-made (3D) titanium plates to standard two titanium mini plates in fixation of mandibular angle fracture.

DETAILED DESCRIPTION:
Eighteen patients with mandibular angle fractures will be selected. In nine fractures, custom-made three dimensional titanium plates will be used for fracture fixation (study group); while in the other nine, conventional two mini plates will be used (control group),via intra oral approach (combined with transbuccal approach) for both groups. Patients will be evaluated clinically, and radiographically (immediate and four months post operative) to evaluate the bone density at the fracture line.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from mandibular angle fracture indicated for open reduction and fixation.
2. Non infected mandibular angle fractures present less than two weeks. 3. Good oral hygiene.

Exclusion Criteria:

1. Medically compromised patients contradicting operation (ASA III, IV & V).
2. Patients receiving radiotherapy or chemotherapy. 3- Bone diseases (Osteoporosis, Osteopetrosis, Osteomalacia…etc.) 4- Pathological fracture. 5- Old untreated fracture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation for the assessment of mean bone density at the fracture line | 4 months
  Mean bone density at the fracture line was assessed using Computed Tomography (CT) scan in Hounsfield Units (HU)

SECONDARY OUTCOMES:
Post operative pain | 3 months
  - Post operative pain This will be subjectively evaluated with a visual analogue scale (VAS) with values from 0 (no pain) to 10 (strongest pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes